CLINICAL TRIAL: NCT06172699
Title: Assert-IQ Insertable Cardiac Monitor Post Market Study
Brief Title: Assert-IQ Implantable Cardiac Monitor (ICM) Post Market Study
Acronym: Assert-IQ
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10468
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation Paroxysmal; Atrial Fibrillation, Persistent; Cardiac Arrhythmia; Ablation
Keywords: atrial fibrillation; Holter monitor; cardiac arrhythmia; arrhythmia risk; syncope; shortness of breath; dizziness; palpitations; tachycardia; sinus pauses; Holter ECG recorder
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Syncope; Dyspnea; Dizziness; Tachycardia | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects successfully implanted with an Abbott Assert-IQ ICM device: Holter monitoring in subjects successfully implanted with an Abbott Assert-IQ ICM device
  Interventions: Device: Holter monitoring in patients who have been successfully implanted with an Abbott Assert-IQ ICM device

INTERVENTIONS:
Device: Holter monitoring in patients who have been successfully implanted with an Abbott Assert-IQ ICM device — All enrolled subjects who meet eligibility criteria will undergo an attempted implant within 30 days of consent. After successful device implant, subjects will be followed at 1 and 12 months. Subjects will be fitted with a Holter monitor during the 1m follow-up visit and will complete a minimum of 72 hours and maximum of up to 7 days of Holter monitoring.

SUMMARY:
This is a prospective, non-randomized, multi-center, real-world post-market study to collect and evaluate data regarding the performance of the enhanced atrial fibrillation detection algorithm of the Assert-IQTM Implantable Cardiac Monitor (ICM) device.

DETAILED DESCRIPTION:
The study's intent is to generate long-term real-world data on the safety, performance, and clinical benefits of the Assert-IQTM ICM device system. This clinical investigation is sponsored by Abbott Medical.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL study inclusion criteria to participate in the study.

1. Have an approved indication AND are scheduled to receive an Assert-IQTM ICM device prior to enrollment in the study.
2. Diagnosed with symptomatic, drug-refractory paroxysmal or persistent AF prior to enrollment in the study and scheduled to undergo a first-time atrial fibrillation ablation.
3. Have a cellular phone or the ability or willing to use a mobile transmitter that is compatible with the myMerlin™ App and able to communicate with the Assert-IQTM ICM device. If a subject doesn't have a cell phone or loses their cell phone, then the site can provide a mobile transmitter to the subject. The study will not provide cell phones.
4. Are 18 years of age or older, or of legal age to give informed consent specific to state and national law.
5. Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

If ANY study exclusion criteria are met, the patient is excluded from the study and cannot be enrolled (recruitment failure).

1. Subject is currently participating in another clinical investigation that could confound the results of this study, without documented pre-approval from Abbott.
2. Subject is implanted with a cardiac implantable electronic device (CIED) with pacing capability.
3. Have a life expectancy of less than 1 year due to any condition.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are diagnosed with symptomatic, drug-refractory paroxysmal or persistent AF, and are scheduled to receive an Assert-IQTM ICM device
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Episode-based AF detection performance metrics | Holter monitor worn by the subjects over a minimum 72-hour and up to 7 days period. An AF episode is defined as AF has greater or equal to 2 minutes (≥2 minutes) in duration.
  Episode-based AF detection performance metrics of the Assert-IQTM ICM device compared to that of simultaneous Holter monitoring in 150 subjects who had received the Assert-IQTM ICM device as part of their standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Kwangdeok Lee, PhD, Study Director — Abbott
Locations (11):
- United States (11):
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Orlando Health, Orlando, Florida
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Trinity Health-Michigan d/b/a Michigan Heart, Ann Arbor, Michigan
  - St. Peter's Health Partners Medical Associates, PC, Albany, New York
  - Trident Medical Center, Charleston, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Shannon Clinic, San Angelo, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Heart Rhythm Associates, The Woodlands, Texas
  - Aurora Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No